CLINICAL TRIAL: NCT03276403
Title: Finding New Criteria for a Revised Primary Graft Dysfunction Score in Lung Transplantation - a Pilot Study
Brief Title: Primary Graft Dysfunction Score in Lung Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assoc.-Prof. Dr. Konrad Hoetzenecker, PhD (Other)
Responsible Party: Sponsor-Investigator, Assoc.-Prof. Dr. Konrad Hoetzenecker, PhD, Assoc.-Prof. Dr. Konraf Hoetzenecker, PhD, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: 1618/2016
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Lung Transplant; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: PiCCO Catheter — The PiCCO Catheter is an investigational device intended to measure lung water content in individuals requiring advanced haemodynamic monitoring. The device system is to be used only in accordance with the approved Investigational Plan on subjects who have signed an informed consent form. Device use is limited to the approved study investigators.

SUMMARY:
The validity of several functional parameters, which could be included in a new PGD scoring system, will be tested in a prospective pilot study of 80 consecutive bilateral lung transplant recipients in high volume lung transplant centers. Functional parameters will be collected at different time points within the first 72hrs after lung transplantation and their accuracy in predicting clinical outcome as well as their correlation with lung water content (measured by PiCCO) will be tested. Insights will serve to generate a hypothesis (a novel PGD score), which can then be tested in future prospective trials.

ELIGIBILITY:
Inclusion Criteria:

* Double lung transplantation for primary pulmonary hypertension (PPH), Fibrosis, cystic fibrosis (CF), Emphysema
* No restrictions regarding donor lungs (marginal donors, EVLP possible)
* No restrictions regarding size reduction (anatomic wedge resections, three lobar, lobar transplantations)

Exclusion Criteria:

* Single-lung transplantation
* Heart-lung transplantation
* Re-transplantation
* Patients with bridge-to-transplantation with a mechanical assist device (extra-corporal membrane oxygenation (v/v, v/a), PA/LA Novalung, ILAactive, ILA)
* Clinical situations leading to inaccurate PiCCO measurements e.g. intracardiac shunts, significant tricuspid regurgitation, cooling
* No access to the femoral artery possible
* Severe postoperative hemorrhage, which leads to hematothorax and makes revision surgery necessary

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving double lung transplantation
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
Primary graft dysfunction | 72 hours after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Hoetzenecker, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (2):
- Medical University of Vienna, Vienna, Austria
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon request